CLINICAL TRIAL: NCT02249234
Title: Randomized Control Trial of the Use of Botox to Treat Chronic Scrotal Pain
Acronym: ROBOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAN-BTX-RCT
Record Dates: First submitted 2014-08-28; First posted 2014-09-25 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Scrotal Pain
Keywords: Scrotal pain; Botox
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Experimental): Botox 200 units reconstituted in 10ml of normal saline for a one-time injection
  Interventions: Drug: Botox
- Saline (Placebo Comparator): Saline 10ml of normal saline for a one-time injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botox
  Other Names: OnabotulinumtoxinA
  Arms: Botox
Drug: Placebo
  Arms: Saline

SUMMARY:
There are no previous reports on the use of OnabotulinumtoxinA (Botox) to treat men with scrotal pain that we found published.

We proposed a pilot study using Botox to block the nerves on a small group of men with chronic scrotal pain (CSP) who have failed the standard medical therapy. The men must have had temporary relief from a testicular cord block using local anaesthetic drug.

The encourage results of the pilot study has given us the background information to proceed with a formal randomised control trial of Botox vs placebo.

We hypothesized that Botox injections to block the testicular nerve will be effective in providing long term pain relief for men with scrotal pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have nociceptive scrotal pain,
* Have no identifiable, reversible causes for the scrotal pain
* Have failed standard medical therapy
* Have responded temporarily to cord blocks

Exclusion Criteria:

* Are interested in trying to conceive with their partners in the next 6 months,
* Have any local infection near the site of the injections,
* Have had an allergic reaction to Botox in the past,
* Are unable to provide informed consent
* Have a history of motor neuron disease or neurogenic bladder
* Who have hemostatic disorder or who are taking aspirin, Coumadin (warfarin), Xarelto (rivaroxaban) or other blood thinners

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Reduction in the visual analog scales for pain | 6 months after entering in trial
  A measure of the change in the visual analog scales for pain.

SECONDARY OUTCOMES:
Reduction in scrotal pain | 6 months after entering in trial
  It will be assessed by the Chronic Epididymitis Symptom Index score.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Jarvi, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada